CLINICAL TRIAL: NCT01872585
Title: Feasibility Study of a Mentalization-based Parenting Program for Female Caregivers Involved in Mental Health Services.
Brief Title: Program for Caregivers Involved With Mental Health Services
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1004006576
Record Dates: First submitted 2012-04-27; First posted 2013-06-07 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Mental Illness
Keywords: Parenting; Mental Illness; Maternal sensitivity; Parent-child relationship
MeSH Terms: conditions — Mental Disorders | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mentalization based therapy (Experimental): Women who are the primary caregivers of a child between the ages of 0-7 years and are involved with mental health services for themselves or a child.
  Interventions: Behavioral: Mentalization based therapy

INTERVENTIONS:
Behavioral: Mentalization based therapy — 12-24 weekly 1 hour individual therapy sessions with Masters level therapists who are trained and supervised by Dr. Suchman (the Principal Investigator) in the Parenting from the Inside Out approach. The broad goals of the program are to help prevent the onset of substance abuse and psychiatric disorders, promote adaptive interpersonal relationships and social-emotional functioning in caregivers and their children, and help prevent the transmission of psychiatric illness across generations

SUMMARY:
The purpose of this two-year pilot study is to adapt a 12-week attachment-based parenting intervention for implementation with female adult caregivers who have or are at risk for long-term interpersonal conflict with family members, children, or significant others and are caring for a child between the ages of birth and 7 years.

DETAILED DESCRIPTION:
The purpose of this two-year pilot study is to adapt a 12-week attachment-based parenting intervention (Parenting from the Inside Out or PIO) originally developed for substance abusing mothers (as part of an ongoing NIDA-funded treatment development study; R01 DA17294) for implementation with female adult caregivers who have or are at risk for long-term interpersonal conflict with family members, children, or significant others and are caring for a child between the ages of birth and 7 years. The PIO intervention involves 12-24 weekly 1 hour individual therapy sessions with Masters level therapists who are trained and supervised by Dr. Suchman (the Principal Investigator) in the PIO approach.

ELIGIBILITY:
Inclusion Criteria:

* receive psychiatric services through the adult or young adult treatment team at the West Haven Mental Health Clinic
* have a child receiving psychiatric services through the child treatment team at the West Haven Mental Health Clinic
* express interest in receiving a parent intervention at the West Haven Mental Health Clinic

Exclusion Criteria:

* severe mental health problems (e.g., suicidal, homicidal, psychosis, thought disorder)
* severely cognitively impaired
* have psychiatric or substance-related symptoms requiring inpatient hospitalization or ambulatory detoxification
* are not fluent in English
* child has a serious illness or significant developmental delay (e.g., cognitive, language, or motor)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maternal reflective functioning | Change at week 12 from baseline
  PDI: Rated on a -1 to +9 scale where a score of 3 indicates simple awareness of mental states, 5 indicates rudimentary recognition of how mental states influence behavior, and above 5 indicates advance rPRFQ-1: Rated on a 7-point scale. 3 subscales: PMM (Pre-mentalizing Mode) with high scores indicating reliance on pre-reflective modes of thinking about child's behavior, NRO (Not Recognizing Opacity) with high scores indicating less recognition of the opaque nature of the child's mental states, and IC (Interest and Curiosity) with high scores indicating more interest and curiosity about the child's underlying mental states.
Maternal reflective functioning | Change at week 24 from baseline
  PDI: Rated on a -1 to +9 scale where a score of 3 indicates simple awareness of mental states, 5 indicates rudimentary recognition of how mental states influence behavior, and above 5 indicates advance rPRFQ-1: Rated on a 7-point scale. 3 subscales: PMM (Pre-mentalizing Mode) with high scores indicating reliance on pre-reflective modes of thinking about child's behavior, NRO (Not Recognizing Opacity) with high scores indicating less recognition of the opaque nature of the child's mental states, and IC (Interest and Curiosity) with high scores indicating more interest and curiosity about the child's underlying mental states.

SECONDARY OUTCOMES:
Coding Interactive Behavior | Change at week 12 from baseline
  The caregiver-child dyad will be given age-appropriate toys and instructed to interact freely and session is videotaped and coded using CIB. Composite scores are scored on a 1 - 5 scale. Composite maternal scales include Sensitivity, Intrusiveness, Limit Setting, and Negative Emotion. Composite Child Scales include Child Involvement, Withdrawal and Compliance. Composite Dyadic Scales include Reciprocity and Dyadic Negative States.
Coding Interactive Behavior | Change at week 24 from baseline
  The caregiver-child dyad will be given age-appropriate toys and instructed to interact freely and session is videotaped and coded using CIB. Composite scores are scored on a 1 - 5 scale. Composite maternal scales include Sensitivity, Intrusiveness, Limit Setting, and Negative Emotion. Composite Child Scales include Child Involvement, Withdrawal and Compliance. Composite Dyadic Scales include Reciprocity and Dyadic Negative States.
Maternal parenting stress | Change at week 12 from baseline
  The PSI yields five scores: Parent Dysfunction, Parent-Child Difficulty, Difficult Child, Defensive Responding, and Total Stress which are standardized to percentile rankings. We will be testing for reduction in each stress domain to below the 85th percentile.
Maternal parenting stress | Change at week 24 from baseline
  The PSI yields five scores: Parent Dysfunction, Parent-Child Difficulty, Difficult Child, Defensive Responding, and Total Stress which are standardized to percentile rankings. We will be testing for reduction in each stress domain to below the 85th percentile.
Maternal depression | Change at week 12 from baseline
  Scores range from 0 to 63. We will be testing for significant reduction in total depression.
Maternal depression | Change at week 24 from baseline
  Scores range from 0 to 63. We will be testing for significant reduction in total depression.
Maternal global psychiatric distress | Change at week 12 from baseline
  The composite Global Severity Index (GSI) from the Brief Symptom Inventory measures current overall symptomatology across multiple domains (e.g., depression, anxiety, interpersonal sensitivity, somatic complaints, paranoid ideation) and has demonstrated good reliability and validity. T scores above 60 on the GSI indicate risk for a clinical disorder.
Maternal global psychiatric distress | Change at week 24 from baseline
  The composite Global Severity Index (GSI) from the Brief Symptom Inventory measures current overall symptomatology across multiple domains (e.g., depression, anxiety, interpersonal sensitivity, somatic complaints, paranoid ideation) and has demonstrated good reliability and validity. T scores above 60 on the GSI indicate risk for a clinical disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Suchman, PhD, Principal Investigator — Yale University
Locations (1):
- West Haven Mental Health Clinic, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Suchman NE, Ordway MR, de Las Heras L, McMahon TJ. Mothering from the Inside Out: results of a pilot study testing a mentalization-based therapy for mothers enrolled in mental health services. Attach Hum Dev. 2016 Dec;18(6):596-617. doi: 10.1080/14616734.2016.1226371. Epub 2016 Aug 30. PMID 27575343